CLINICAL TRIAL: NCT06388603
Title: A National, Prospective, Randomized, Multicenter, Controlled Comparison of Bioactive Glass S53P4 Versus Standard of Care Treatment of Diabetic Foot Osteomyelitis in the Forefoot
Brief Title: RCT on Bioactive Glass S53P4 in Diabetic Foot Osteomyelitis in the Forefoot (DFORCT)
Acronym: DFORCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Ovest Milanese (Other)
Collaborators: Hippocrates Research (Other); Bonalive Biomaterials Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFORCT012023
Record Dates: First submitted 2024-04-19; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Osteomyelitis - Foot
Keywords: Diabetic Foot; Osteomyelitis; Forefoot
MeSH Terms: conditions — Diabetic Foot; Osteomyelitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care - Osteomyelitis treatment (Active Comparator): Subjects randomized in this group will be treated according to standard of care for the surgical managment of Osteomyelitis in the forefoot in patient suffering from diabetic foot syndrome. All standard of care approaches will be allowed (e.g use of bone sobsitutes, cements, cements loaded with antibiotics etc) with the only exception of Bioactive Glasses.
  Interventions: Other: Standard of Care
- Bioactive Glass (Experimental): Subjects randomized in this group will be treated using the S53P4 Bioactive Glass of Bonalive Biomaterials Ltd; in the form of:
  * Bonalive Granules 2.5 CC (0.5-0.8 MM)
  * Bonalive Putty 2.5 CC (SIRINGA 0.5-0.8 MM)
  The quantity that will be implanted will vary according to the bone cavity of each patient.
  Interventions: Device: Bioactive Glass

INTERVENTIONS:
Device: Bioactive Glass — Bonalive Granules and Bonalive Putty will be used (according to their IFU and CE certification) to fill the bone void after the debridment of infected tissue as they have osteoconductive and osteostimulative properties that allow bone rigeneration. Moreover, Bonalive Granules also present some bacteria growth inhibiting properties to combact bone infection propoer of Ostemyelitis.
  Other Names: Bonalive Granules RDM: 856052; manufacturer code:13120; Bonalive Putty RDM: 855194; manufacturer code:16120
  Arms: Bioactive Glass
Other: Standard of Care — The investigators are left free to proceed according to the normal standar procedure they normally use. The procedures can vary according to investigator judgment also depending on the state of Osteomylitis.
  Arms: Standard of Care - Osteomyelitis treatment

SUMMARY:
The Study will be a prospective multicenter randomized trial, focused on the management of acute and chronic Osteomilytis in Diabetic Foot patients. The aim of this Study will be to compare the effectiveness and safety of S53P4 bioactive glass, medical device class III used as per its CE mark indication and Instruction For Use, in the surgical management of OM in the forefoot performed as per local surgical standard of care, in the same indications in a group of Diabetic Foot patients admitted in highly specialized dedicated centers.

Participants will randomized into two groups:

* Patients in Group A will be treated with surgical removal of the affected bone, debridement of infected soft tissues and systemic antibiotic therapy targeted on the sampling on the bone during the surgical procedure, with or without use of bone substitutes (with the only exception of Bioactive glasses) according to the judgement of the operator as per normal practice.
* Patients in Group B will be debrided as well and the infected bone will be debrided without eliminating completely the structure of the bone, but instead preserving the cortex, while all the soft bone visibly infected will be removed and then replaced with Bioactive glass, as per IFU, (S53P4 - Bonalive® granules and putty, Bonalive Biomaterials Ltd. Finland) and then closed for primary intention whenever possible.

DETAILED DESCRIPTION:
Patient with a diagnosis of ostemileytis localised in the forefoot will be randomized into two groups.

* Patients in Group A will be treated with surgical removal of the affected bone, debridement of infected soft tissues and systemic antibiotic therapy targeted on the sampling on the bone during the surgical procedure, with or without use of bone substitutes (with the only exception of Bioactive glasses) according to the judgement of the operator as per normal practice.
* Patients in Group B will be debrided as well and the infected bone will be debrided without eliminating completely the structure of the bone, but instead preserving the cortex, while all the soft bone visibly infected will be removed and then replaced with Bioactive glass, as per IFU, (S53P4 - Bonalive® granules and putty, Bonalive Biomaterials Ltd. Finland) and then closed for primary intention whenever possible.

In any case a primary intent closure is pursued, both in Group A and B, a vacuum percutaneous drainage would be placed before closing the wound and removed in 2nd post-operative day, if necessary, by the surgeon.

Systemic antibiotic therapy will be started immediately on empirical basis, as per normal practice.

After the removal of drainage, or after the first post-operative control in 2nd post-operative day, as done routinely at study sites, patients will be evaluated biweekly either if they are still admitted or if they were dismissed and will be followed up by investigators blinded toward the groups.

At each visit local conditions and eventual dressing changes will be recorded, alongside with any possible complication, like non-healing, re-infection, and any systemic and local adverse event.

Patients will be followed every second week up to 3 months or until complete healing and then at six months and 12 months from surgical interventions. At six-month and 12 -month follow-up, rate of healing and recurrences will be checked; x-rays will be performed at pre-operation visit, immediate post and at 12 months Follow Up visit. Histopathological samples collected as per normal practice during the surgery will be analyzed with standard protocol in local laboratories. Healing will be defined as complete re-epithelization of the lesion, without secretion or drainage, confirmed at two successive follow-up visits. For the sake of calculating healing time, healing will be attributed to the first visit. At each visits a local and systemic evaluation of the wound will be done as per normal practice. A photo of the wound will be taken at visits: Pre-operative , Immediate post-op, 6 weeks post-op, 6 months and 12 months after the surgical procedure. Laboratory exams will be performed as per hospital standard of care. At pre-operative and 6 months and 12 months visits patients compile Quality of Life and Foot Function Index Questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained.
2. Male or female patients >= of 18 years old.
3. They should have type I since at least 5 years or type II DM
4. They should have a diagnosis - confirmed by imaging and culture - of OM localized in the forefoot not responding for at least 2 up to 6 weeks to systemic antibiotic therapy and/or associated with soft tissue infection, abscess, phlegmon, necrosis, and for which a surgical debridement is indicated.
5. They should have palpable pulses on TP or DP at the ankle in the affected limb, and/or ABPI >0.7 and <1.2 and /or TcPO2 at dorsum of the foot ≥36 mmHg.
6. They should be able to accomplish with the procedures and prescriptions indicated by the Study protocol, particularly with the offloading prescription, as well as they should be willing and able to attend and respect the program of control visits and medications.
7. Anatomical area: forefoot.

Exclusion Criteria:

1. They should not have metabolic decompensation as witnessed by HbA1c >109 mmol/mol (> 12%).
2. They should not have major amputation on the contra-lateral limb.
3. They should not have acute or chronic Charcot's foot in the affected foot.
4. They should not have undergone surgical or endovascular revascularization in the affected foot in the month preceding the enrollment.
5. They should not be taking corticosteroids, bisphosphonates, immunosuppressants, and more in general any drug which might interfere with bone metabolism or tissue repair, in thejudgment of investigators.
6. They should not have ESRD in dialysis.
7. They should not be bedridden or not ambulating.
8. They should not have a life expectancy shorter than one year.
9. They should not be too ill to sustain a surgical procedure under loco-regional anesthesia.
10. They should not have severe disease which might interfere with the expected course of the disease and therapy.
11. Hypersensitivity to any product ingredient(s) or history of anaphylactic reactions.
12. Participation in another interventional studies within 45 days prior to the start of the present study.
13. Predictable poor compliance or inability to communicate well with the investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
healing rate | 6-month
  complete re-epithelization of the lesion, without secretion or drainage, confirmed at two successive follow-up visits.

SECONDARY OUTCOMES:
Duration of antibiotic therapy | through study completion, an average of 1 year
  systemic antibiotic therapy will be prescribed after intervention and its duration can vary according to infection state.
Rate of recurrences | 6-months and 12-month
  After intervention bone infections proper of osteomyelitis can recur
Number of re-interventions because of the same lesion | through study completion, an average of 1 year
  If an infection recur might be necessery to procede with a re-intervention.
Timing of re-interventions because of the same lesion | through study completion, an average of 1 year
  If an infection recur might be necessery to procede with a re-intervention.
Proportion of patients undergoing amputations | through study completion, an average of 1 year
  In same severe cases minor or major amputations can be neccessary
Patients' Quality of Life | 6-months and 12-month
  The quality of life of patient will be evaluated using EQ-5D-5L from 0 (worse) to 100 (better)
Patients' Quality of Life | 6-months and 12-month
  The quality of life of patient will be evaluated with Foot Function Index from 0 (better) to 170 (worse)
Time back to walk | through study completion, an average of 1 year
  It will be registered when patients can go back to walk aftern the intervention
Characteristics of surgery | intra-operative
  data about characteristics (type) of surgeries will be collected
Length of surgery | intra-operative
  data about the lenght (timing) of surgeries will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Roberto De Giglio, Med Doctor, Principal Investigator — ASST Ovest Milanese
Locations (7):
- Italy (7):
  - ASUGI Azienda Sanitaria Universitaria Giuliano Isontina - Ospedale Monfalcone, Monfalcone, Gorizia
  - ASST Ovest Milanese - Ospedale di Abbiategrasso, Abbiategrasso, Milano
  - Casa di Cura Abano Terme - POLICLINICO ABANO TERME, Abano Terme, Padova
  - USL Sud Est Toscana - Ospedale San Donato, Arezzo
  - AUSL Romagna - Ospedale Morgagni Pierantoni, Forlì
  - Azienda USL Toscana Nord Ovest - Ospedale Campo di Marte, Lucca
  - AOU Pisana - Ospedale di Cisanello, Pisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Giglio R, Di Vieste G, Mondello T, Balduzzi G, Masserini B, Formenti I, Lodigiani S, Pallavicini D, Pintaudi B, Mazzone A. Efficacy and Safety of Bioactive Glass S53P4 as a Treatment for Diabetic Foot Osteomyelitis. J Foot Ankle Surg. 2021 Mar-Apr;60(2):292-296. doi: 10.1053/j.jfas.2020.06.029. Epub 2020 Sep 6. PMID 33358382
- [Background] Prompers L, Huijberts M, Apelqvist J, Jude E, Piaggesi A, Bakker K, Edmonds M, Holstein P, Jirkovska A, Mauricio D, Ragnarson Tennvall G, Reike H, Spraul M, Uccioli L, Urbancic V, Van Acker K, van Baal J, van Merode F, Schaper N. High prevalence of ischaemia, infection and serious comorbidity in patients with diabetic foot disease in Europe. Baseline results from the Eurodiale study. Diabetologia. 2007 Jan;50(1):18-25. doi: 10.1007/s00125-006-0491-1. Epub 2006 Nov 9. PMID 17093942
- [Background] Prompers L, Huijberts M, Apelqvist J, Jude E, Piaggesi A, Bakker K, Edmonds M, Holstein P, Jirkovska A, Mauricio D, Tennvall GR, Reike H, Spraul M, Uccioli L, Urbancic V, Van Acker K, Van Baal J, Van Merode F, Schaper N. Delivery of care to diabetic patients with foot ulcers in daily practice: results of the Eurodiale Study, a prospective cohort study. Diabet Med. 2008 Jun;25(6):700-7. doi: 10.1111/j.1464-5491.2008.02445.x. PMID 18544108
- [Background] Lipsky BA, Aragon-Sanchez J, Diggle M, Embil J, Kono S, Lavery L, Senneville E, Urbancic-Rovan V, Van Asten S; International Working Group on the Diabetic Foot; Peters EJ. IWGDF guidance on the diagnosis and management of foot infections in persons with diabetes. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:45-74. doi: 10.1002/dmrr.2699. No abstract available. PMID 26386266
- [Background] Lalidou F, Kolios G, Drosos GI. Bone infections and bone graft substitutes for local antibiotic therapy. Surg Technol Int. 2014 Mar;24:353-62. PMID 24504740
- [Background] Hanssen AD. Local antibiotic delivery vehicles in the treatment of musculoskeletal infection. Clin Orthop Relat Res. 2005 Aug;(437):91-6. doi: 10.1097/01.blo.0000175713.30506.77. PMID 16056032
- [Background] Vatan A, Saltoglu N, Yemisen M, Balkan II, Surme S, Demiray T, Mete B, Tabak F; Study Group, Cerrahpasa Diabetic Foot. Association between biofilm and multi/extensive drug resistance in diabetic foot infection. Int J Clin Pract. 2018 Mar;72(3):e13060. doi: 10.1111/ijcp.13060. Epub 2018 Jan 30. PMID 29381248
- [Background] Lindfors NC, Hyvonen P, Nyyssonen M, Kirjavainen M, Kankare J, Gullichsen E, Salo J. Bioactive glass S53P4 as bone graft substitute in treatment of osteomyelitis. Bone. 2010 Aug;47(2):212-8. doi: 10.1016/j.bone.2010.05.030. PMID 20624692
- [Background] Peltola M, Aitasalo K, Suonpaa J, Varpula M, Yli-Urpo A. Bioactive glass S53P4 in frontal sinus obliteration: a long-term clinical experience. Head Neck. 2006 Sep;28(9):834-41. doi: 10.1002/hed.20436. PMID 16823870
- [Background] McAndrew J, Efrimescu C, Sheehan E, Niall D. Through the looking glass; bioactive glass S53P4 (BonAlive(R)) in the treatment of chronic osteomyelitis. Ir J Med Sci. 2013 Sep;182(3):509-11. doi: 10.1007/s11845-012-0895-5. Epub 2013 Jan 5. PMID 23292733
- [Background] Piaggesi A, Goretti C, Iacopi E, Clerici G, Romagnoli F, Toscanella F, Vermigli C. Comparison of Removable and Irremovable Walking Boot to Total Contact Casting in Offloading the Neuropathic Diabetic Foot Ulceration. Foot Ankle Int. 2016 Aug;37(8):855-61. doi: 10.1177/1071100716643429. Epub 2016 Apr 15. PMID 27083507
- [Background] Kastrin M, Urbancic Rovan V, Frangez I. Possible Advantages of S53P4 Bioactive Glass in the Treatment of Septic Osteoarthritis of the First Metatarsophalangeal Joint in the Diabetic Foot. J Clin Med. 2021 Mar 15;10(6):1208. doi: 10.3390/jcm10061208. PMID 33803930
- [Background] Iacopi E, Pieruzzi L, Goretti C, Piaggesi A. Pilot Experience on the Use of S53P4 Bioactive Glass in the Surgical Management of Diabetic Foot Osteomyelitis. Int J Low Extrem Wounds. 2022 Mar;21(1):57-64. doi: 10.1177/1534734620926003. Epub 2020 Jun 8. PMID 32506987
- [Background] Munukka E, Lepparanta O, Korkeamaki M, Vaahtio M, Peltola T, Zhang D, Hupa L, Ylanen H, Salonen JI, Viljanen MK, Eerola E. Bactericidal effects of bioactive glasses on clinically important aerobic bacteria. J Mater Sci Mater Med. 2008 Jan;19(1):27-32. doi: 10.1007/s10856-007-3143-1. Epub 2007 Jun 14. PMID 17569007